CLINICAL TRIAL: NCT06250075
Title: Effects of the Use of Probiotics on the Intestinal Microbiota, Clinical-Nutritional and Immunological Status of Patients Gastrectomized for Gastric Cancer: A Randomized Clinical Trial
Brief Title: Effects of the Use of Probiotics on the Intestinal Microbiota of Patients With Gastric Cancer
Acronym: PRONIC-G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Amazonas (Other)
Responsible Party: Principal Investigator, Abner Souza Paz, RD, Principal Investigator, Universidade Federal do Amazonas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6.014.436
Record Dates: First submitted 2024-01-05; First posted 2024-02-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Gastric Adenocarcinoma; Gastric Cancer; Microbiome; Cytokines; Nutritional Status
Keywords: Gastric Cancer; Microbiome; Nutritional Status; Cytokines
MeSH Terms: conditions — Stomach Neoplasms | interventions — Dosage Forms; Probiotics; Methods

STUDY DESIGN:
Intervention Model Description: In time 1 of the research, patients will be distributed through the Randomizer Clinical Trial Lite application into 4 groups (G1, G2, G4 and G5) to receive 1 capsule a day of probiotics (groups G1 and G4) will receive a formulation containing 20 billion of microorganisms. In group G2 (no intervention), treatment with standard nutrition, without the use of probiotics. The intervention product (probiotic capsules) will be distributed and packaged according to randomization for blinding. In the case of group G3 (control), they will receive probiotic capsules after the end of groups G1 and G2. Both groups that will use probiotic capsules, 1 capsule per day, in the same shift, must continue for 7 days, without interruption in monitoring. In relation to groups G4 and G5, they constitute time 2 of the research, with G4 being the group that will use probiotics following the G1 standard and G5 will use placebo capsules with 0.5g of calcium carbonate to test the power of the intervention.
Who Masked: Participant
Masking Description: For the first stage of the research, patients eligible for cancer gastrectomies were invited at FCECON on an outpatient basis or through the surgical map on the day of admission. Randomization took place through a specific application called Randomizer for Clinical Trial Lite. Different wards were assigned to each group to avoid contact between research participants (G1 intervention and G2 non-intervention). For the G3 (control) group, they will be recruited by invitation, they must be FCECON employees, this group will specifically be matched by the socioeconomic level of the patients in the G1 group. The G4 and G5 groups will be recruited and randomized in the second stage of the research after the end of the collection of the G1 and G2 groups, for analysis of clinical outcomes in the 7-day postoperative period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- G1 Intervention Group (Experimental): In group 1, the intervention will take place with intake from the 1st day Post-OP when releasing the diet (Orally or ENT) and up to 7 days post-operatively with probiotic capsules.
  Interventions: Dietary Supplement: Formulation with probiotics
- Non-Intervention Group G2 (No Intervention): Group G2 followed general nutritional guidelines. This group will not take probiotics, it will be the surgical comparator.
- G3 Negative Control Group (Sham Comparator): Group G3 (guest employees) will follow the intake of probiotic capsules for 7 days during follow-up, without surgical intervention, these will be chosen at random and standardized by social level paired with G1
  Interventions: Dietary Supplement: Formulation with probiotics
- Intervention for Clinical Outcomes -G4 (Active Comparator): The G4 and G5 groups will be recruited and randomized in the second stage of the research after the end of the collection of the G1 and G2 groups, for analysis of clinical outcomes in the 7-day postoperative period.
  Interventions: Dietary Supplement: Formulation with probiotics
- Non-intervention for Clinical Outcomes -G5 (Placebo Comparator): G5 will use placebo capsules with 0.5g calcium carbonate to test the power of the intervention in reducing postoperative surgical complications or not.
  Interventions: Other: Non-intervention for Clinical Outcomes -G5

INTERVENTIONS:
Dietary Supplement: Formulation with probiotics — Lactobacillus acidophilus NCFM®, Lactobacillus paracasei Lpc-37 ™, Bifidobacterium lactis Bi-04™, Bifidobacterium lactis Bi-07™, Bifidobacterium bifidum Bb-02™)
  Other Names: G1 Intervention Group; G3 Negative Control Group; Intervention for Clinical Outcomes -G4
  Arms: G1 Intervention Group; G3 Negative Control Group; Intervention for Clinical Outcomes -G4
Other: Non-intervention for Clinical Outcomes -G5 — only observation of clinical outcomes in the postoperative period
  Other Names: Non-intervention
  Arms: Non-intervention for Clinical Outcomes -G5

SUMMARY:
The objective of this randomized controlled, prospective clinical study, composed of 5 groups, G1, G2, G3, G4 and G5 is [Evaluate the intestinal microbiota profile, nutritional, immunological status and inflammatory profile, before and after total or partial removal surgery (gastrectomies) for gastric cancer, in a patient using probiotic supplements.] The main questions it aims to answer are:

* probiotics are capable of modulating the immune response and microbiota in cancer patients who will undergo surgery
* surgery itself alters the immunological pattern and microbiota of cancer patients Participants will be divided into groups for evaluation and the G1 intervention group will take probiotic capsules.

The researchers will compare groups G1, G2 with G3 (negative control group) to see if there are differences between using probiotics or not, in controlling the immune response and if there are significant changes in their intestinal microbiota. Groups G4 and G5 will also be compared, where in these we will only measure the power of the use of probiotics in reducing surgical complications in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for total or partial gastrectomy;
* Ages from 18 years old.

Exclusion Criteria:

* Palliative patients
* Use of probiotics and prebiotics in the last 15 days;
* Patients who are unable to complete all monitoring steps;
* AIDS patients;
* Diabetic patients;
* Pregnant patients;
* Patients with Autoimmune Diseases;
* Patients with Liver Diseases;
* Patients with Kidney Disease;
* Patients with Inflammatory Bowel Diseases.
* Patients who have MCP (pacemaker),
* Patients with severe Edema,
* Patients with titanium plates in any limb of the body
* Patients who for some reason had their surgeries suspended during follow-up.
* Patients undergoing mechanical colon preparation in the last 30 days.
* Patients not resident/domiciled in Amazonas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Modulation of the Immune Response | twelve months
  We will measure (measure the concentration) of inflammatory cytokines through flow cytometry, and then observe whether the intervention interferes negatively or positively in the inflammatory pattern.
Modulation of the Intestinal Microbiota | twelve months
  The use of probiotics positively interfered in maintaining a change in the pre-surgical microbial profile, in relation to the post-surgical one.
The use of probiotics can modify the incidence of postoperative complications | twelve months
  During surgery, many inflammatory factors can interfere with the appearance of postoperative complications. We assume that the use of probiotics can beneficially modulate surgical complications.

SECONDARY OUTCOMES:
Modulation of nutritional parameters with the use of probiotics-weight and height | twelve months
  Nutritional measurements such as weight and height will be combined to obtain BMI and evaluate body mass, as biological markers that can be modulated with the use of probiotics.
Modulation of nutritional parameters using probiotics-phase angle | twelve months
  Nutritional measurements such as phase angle (a measurement obtained by applying electrical bioimpendance, as a biological marker that can be modulated with the use of probiotics

CONTACTS AND LOCATIONS:
Locations (1):
- Abner Souza Paz, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: Undecided